CLINICAL TRIAL: NCT00608426
Title: Proactive Tobacco Treatment for Diverse Veteran Smokers
Brief Title: Proactive Tobacco Treatment for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IAB 05-303
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Smoking Cessation; Smoking Tobacco
Keywords: African Americans; telephone counseling; community health planning; ethnic groups
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Group who can elect to receive reactive (usual) care for smoking cessation.
- Proactive Care (Experimental): Group who will be proactively offered smoking cessation care with their choice of smoking cessation services (telephone care or in-person care).
  Interventions: Behavioral: Proactive Outreach with choice of telephone or in-person smoking cessation services

INTERVENTIONS:
Behavioral: Proactive Outreach with choice of telephone or in-person smoking cessation services — This group of participants is sent a recruitment letter, then receives a phone call to offer them their choice of smoking cessation services (either telephone care or in-person care).
  Arms: Proactive Care

SUMMARY:
Tobacco use is the leading cause of premature death in the United States and disproportionately affects Veterans and certain racial/ethnic minority groups. Most smokers are interested in quitting; however, current tobacco use treatment approaches are reactive and require smokers to initiate treatment or depend on the provider to initiate smoking cessation care. As a result, most smokers do not receive comprehensive, evidence-based treatment for tobacco use that includes intensive behavioral counseling along with pharmacotherapy. Proactive tobacco treatment integrates population-based treatment (i.e., proactive outreach) and individual-level treatment (i.e., smoking cessation counseling and pharmacotherapy) to address both patient and provider barriers to comprehensive care.

DETAILED DESCRIPTION:
1. BACKGROUND/RATIONALE Tobacco use remains the number one cause of premature death and morbidity in the United States. Most cigarette smokers want to quit smoking, and about 50% make a quit attempt each year, but only 6% achieve long-term cessation. This randomized controlled trial - the Veterans Victory over Tobacco Study - compared the effects of a proactive tobacco cessation care model versus a traditional cessation care model on the use of tobacco treatment and subsequent population-level smoking cessation rates. Veterans from four VAMCs were recruited from 10/09 to 9/10 and were randomized to either usual care (i.e., reactive care) or the proactive care intervention. Veterans in the usual care group (n=2,604) received access to tobacco treatment services from their VAMC. Veterans in the proactive care intervention group (n=2,519) received proactive outreach (mailed invitation materials followed by telephone outreach); and were offered a choice of smoking cessation services (telephone care or in-person care). The primary outcome was six-month prolonged smoking abstinence one year after randomization. Investigators also analyzed baseline demographics, clinical characteristics (i.e., distance to VAMC, comorbid psychiatric conditions), and smoking history.
2. OBJECTIVES The primary objectives of this study were to (1) Assess the effect of a proactive care intervention on population-level smoking abstinence rates (i.e., abstinence among all smokers including those who use and do not use treatment) and on use of evidence-based tobacco treatments compared to reactive/usual care among a diverse population of Veteran smokers, (2) Compare the effect of proactive care on population-level smoking abstinence rates and use of tobacco treatments between African American and White smokers, and (3) Determine the cost-effectiveness of the proactive care intervention.
3. METHODS In this prospective randomized controlled trial, we identified a population-based registry of current smokers (N=6400) from four Department of Veterans Affairs (VA) Medical Centers facilities using the VA electronic medical record, who were randomized to proactive care or usual care. The proactive care intervention combines: (1) proactive outreach and (2) offer of choice of smoking cessation services (telephone or face-to-face). Proactive outreach included mailed invitations followed by telephone outreach with motivational enhancement (up to 6 call attempts) to encourage smokers to seek treatment with choice of services. Proactive care participants who chose telephone care received VA telephone counseling and access to pharmacotherapy. Proactive care participants who chose face-to-face care were referred to their VA facility's smoking cessation clinic. Usual care group participants had access to standard smoking cessation services provided by their VA facility and their VA primary care provider. Usual care participants could also call their local state telephone quitline. Because this study was testing proactive outreach, smokers were randomized prior to contact and a baseline survey was administered after randomization using a multiple-wave mailed questionnaire protocol. Additional baseline data were extracted from VA administrative databases. Outcomes from both groups were collected 12 months post-randomization from participant surveys and from VA administrative databases. The primary outcome was population-level cessation at one year using a self-reported, 6-month prolonged smoking abstinence measure.
4. STATUS We have successfully conducted a multi-site population-based randomized controlled trial. Our primary outcomes paper was published by the JAMA Internal Medicine online in March 2014 and we are currently working on a second manuscript.
5. CLINICAL SIGNIFICANCE In this study, we tested a proactive care intervention that harnesses the power of the electronic medical record to identify populations of smokers in a health care system and capitalize on the availability of validated telephone care protocols to efficiently deliver intensive behavioral counseling and facilitate access to pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker, identified by tobacco use clinical reminder.

Exclusion Criteria:

* ICD-9 diagnosis of dementia (290.xx or 331.xx).
* Greater than 10 VA mental health clinic visits in past 12 months.
* Missing phone number or mailing address.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6400 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven S. Fu, MD MSCE, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (5):
- United States (5):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Fu SS, van Ryn M, Sherman SE, Burgess DJ, Noorbaloochi S, Clothier B, Joseph AM. Population-based tobacco treatment: study design of a randomized controlled trial. BMC Public Health. 2012 Mar 6;12:159. doi: 10.1186/1471-2458-12-159. PMID 22394386
- [Result] Fu SS, van Ryn M, Sherman SE, Burgess DJ, Noorbaloochi S, Clothier B, Taylor BC, Schlede CM, Burke RS, Joseph AM. Proactive tobacco treatment and population-level cessation: a pragmatic randomized clinical trial. JAMA Intern Med. 2014 May;174(5):671-7. doi: 10.1001/jamainternmed.2014.177. PMID 24615217
- [Result] Burgess DJ, van Ryn M, Noorbaloochi S, Clothier B, Taylor BC, Sherman S, Joseph AM, Fu SS. Smoking cessation among African American and white smokers in the Veterans Affairs health care system. Am J Public Health. 2014 Sep;104 Suppl 4(Suppl 4):S580-7. doi: 10.2105/AJPH.2014.302023. PMID 25100424
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Danan ER, Sherman SE, Clothier BA, Burgess DJ, Pinsker EA, Joseph AM, Noorbaloochi S, Fu SS. Smoking Cessation among Female and Male Veterans before and after a Randomized Trial of Proactive Outreach. Womens Health Issues. 2019 Jun 25;29 Suppl 1(Suppl 1):S15-S23. doi: 10.1016/j.whi.2019.04.001. PMID 31253237
- [Derived] Danan ER, Fu SS, Clothier BA, Noorbaloochi S, Hammett PJ, Widome R, Burgess DJ. The Equity Impact of Proactive Outreach to Smokers: Analysis of a Randomized Trial. Am J Prev Med. 2018 Oct;55(4):506-516. doi: 10.1016/j.amepre.2018.05.023. Epub 2018 Aug 20. PMID 30139707
- [Derived] Melzer AC, Pinsker EA, Clothier B, Noorbaloochi S, Burgess DJ, Danan ER, Fu SS. Validating the use of veterans affairs tobacco health factors for assessing change in smoking status: accuracy, availability, and approach. BMC Med Res Methodol. 2018 May 11;18(1):39. doi: 10.1186/s12874-018-0501-2. PMID 29751746
- [Derived] Japuntich SJ, Sherman SE, Joseph AM, Clothier B, Noorbaloochi S, Danan E, Burgess D, Rogers E, Fu SS. Proactive tobacco treatment for individuals with and without a mental health diagnosis: Secondary analysis of a pragmatic randomized controlled trial. Addict Behav. 2018 Jan;76:15-19. doi: 10.1016/j.addbeh.2017.07.024. Epub 2017 Jul 15. PMID 28735036
- [Derived] Danan ER, Joseph AM, Sherman SE, Burgess DJ, Noorbaloochi S, Clothier B, Japuntich SJ, Taylor BC, Fu SS. Does Motivation Matter? Analysis of a Randomized Trial of Proactive Outreach to VA Smokers. J Gen Intern Med. 2016 Aug;31(8):878-87. doi: 10.1007/s11606-016-3687-1. Epub 2016 Apr 12. PMID 27071399

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the time of the baseline survey, 1277 subjects were excluded for not meeting eligiblitiy criteria: 428 declined to participate; 201 were misclassfied as cigarette smokers (never used cigarettes or smokeless tobacco user); 444 were former smokers (rather than current smokers); 179 had incorrect mailing addresses; and 25 were deceased.
Period: Overall Study
Arm/Group | Usual Care | Proactive Care
Started | 2604 | 2519
Completed | 1768 (This is total # of completed surveys. Not completed primary outcome.) | 1614 (This is total # of completed surveys. Not completed primary outcome.)
Not Completed | 836 | 905
Not completed — Death | 32 | 36
Not completed — Lost to Follow-up | 485 | 521
Not completed — refused, health issues, wrong address | 319 | 348

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Proactive Care | Total
Number analyzed (Participants) | 2604 | 2519 | 5123
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.2) | 55.8 (15.1) | 56.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 141 | 299
  Male | 2446 | 2378 | 4824
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1713 | 1603 | 3316
  Black | 568 | 595 | 1163
  Hispanic | 120 | 111 | 231
  Other | 203 | 210 | 413
Married [Number; unit: participants]
  Married | 1156 | 1108 | 2264
  Not Married | 1448 | 1411 | 2859
Distance to the VA hospital, miles [Number; unit: participants]
  <5 | 212 | 174 | 386
  5-10 | 472 | 456 | 928
  >10-25 | 698 | 662 | 1360
  >25-50 | 425 | 436 | 861
  >50 | 797 | 791 | 1588
Smoking related cancer [Number; unit: participants]
  Cancer | 57 | 71 | 128
  No cancer | 2547 | 2448 | 4995
Smoking related cardiovascular disease [Number; unit: participants]
  Yes | 703 | 677 | 1380
  No | 1901 | 1842 | 3743
Smoking related respiratory disease [Number; unit: participants]
  Yes | 500 | 458 | 958
  No | 2104 | 2061 | 4165
Presence of psychiatric co-morbidity [Number; unit: participants]
  None | 1383 | 1335 | 2718
  One | 612 | 605 | 1217
  Two or more | 609 | 579 | 1188
Depression [Number; unit: participants]
  Yes | 565 | 552 | 1117
  No | 2039 | 1967 | 4006
Anxiety Disorder [Number; unit: participants]
  Yes | 247 | 289 | 536
  No | 2357 | 2230 | 4587
Post-traumatic stress disorder [Number; unit: participants]
  Yes | 216 | 216 | 432
  No | 2388 | 2303 | 4691
Serious mental illness [Number; unit: participants]
  Yes | 177 | 161 | 338
  No | 2427 | 2358 | 4785
Other psychiatric disorder [Number; unit: participants]
  Yes | 430 | 416 | 846
  No | 2174 | 2103 | 4277
Other substance use disorder [Number; unit: participants]
  Yes | 534 | 481 | 1015
  No | 2070 | 2038 | 4108

OUTCOME MEASURES:

1. Primary Outcome: Self-reported, Smoking Abstinence Rate: 6-month Prolonged Abstinence
Time Frame: 12 months after randomization
Population: Out of the 3382 completed follow-up surveys, 3307 completed the primary smoking-abstinence outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Proactive Care
Number analyzed (Participants) | 1734 | 1573
percentage of participants | 10.9 | 13.5
Statistical Analysis 1: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = .02, Regression, Logistic

2. Secondary Outcome: Treatment Utilization Rates for Counseling and/or Pharmacotherapy
Time Frame: 12 months after randomization
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Proactive Care
Number analyzed (Participants) | 1734 | 1573
percentage of participants
  Telephone counseling | 2.2 | 12.7
  In-person counseling | 6 | 5.5
  Used medication | 39 | 41.1
  Combination counseling and medication | 5.1 | 12.8
  Attended VA smoking cessation clinic | 3.4 | 3.2
  Received VA smoking cessation medication | 29.5 | 34.5
Statistical Analysis 1: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p < .001, Mixed effects logistic regression — for the comparison of telephone counseling between the two groups
Statistical Analysis 2: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = 0.57, Mixed effects logistic regression — for the comparison of in-person counseling between the two groups
Statistical Analysis 3: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = .15, Mixed effects logistic regression — for the comparison of used medications between the two groups
Statistical Analysis 4: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p < .001, Mixed effects logistic regression — for the comparison of combination counseling and medication between the two groups
Statistical Analysis 5: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = .77, Mixed effects logistic regression — for the comparison of attended VA smoking cessation clinic between the two groups
Statistical Analysis 6: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = .002, Mixed effects logistic regression — for the comparison of received VA smoking cessation medication between the two groups

3. Secondary Outcome: 7-day Point Prevalence Abstinence
Time Frame: 12 months after randomizatoin
Population: Out of the 3382 completed follow-up surveys, 3056 completed the 7-day point prevalence outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Proactive Care
Number analyzed (Participants) | 1603 | 1453
percentage of participants | 15.1 | 17.1
Statistical Analysis 1: Comparison: Usual Care vs Proactive Care; Test type: Superiority or Other; p = 0.13, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Usual Care | Proactive Care
Serious Adverse Events (participants affected / at risk) | 0/2604 | 0/2519
Other Adverse Events (participants affected / at risk) | 0/2604 | 0/2519

LIMITATIONS AND CAVEATS:
Smoking abstinence rates were not biochemically verified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No